CLINICAL TRIAL: NCT01984775
Title: An Evaluator-Blinded Study to Evaluate the Cumulative Irritation Potential of Topically-Applied GSK2894512 Cream in Healthy Subjects
Brief Title: A Study to Evaluate the Irritation Potential of GSK2894512 Cream on Skin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 117191
Record Dates: First submitted 2013-10-31; First posted 2013-11-15 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Psoriasis
Keywords: safety; dermal; GSK2894512; Cumulative irritation
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- GSK2894512 0.5% (Experimental): Each subject will receive a topical application of GSK2894512 0.5% under semi-occlusive patch conditions once daily (OD) for 21 days.
  Interventions: Drug: GSK2894512 cream
- GSK2894512 1% (Experimental): Each subject will receive a topical application of GSK2894512 1% under semi- occlusive patch conditions OD for 21 days.
  Interventions: Drug: GSK2894512 cream
- GSK2894512 2% (Experimental): Each subject will receive a topical application of GSK2894512 2% under semi-occlusive patch conditions OD for 21 days.
  Interventions: Drug: GSK2894512 cream
- Vehicle (Placebo Comparator): Each subject will receive a topical application of Vehicle cream under semi-occlusive patch conditions OD for 21 days.
  Interventions: Drug: Vehicle cream
- Sodium lauryl sulfate 0.1% (Active Comparator): Each subject will receive a topical application of 0.2 milliliter (mL) of Sodium lauryl sulfate under semi-occlusive patch conditions OD for 21 days. This will serve as a positive control.
  Interventions: Drug: Positive control
- Petrolatum (Active Comparator): Each subject will receive a topical application of 0.2 mL of Petrolatum under semi-occlusive patch conditions OD for 21 days. This will serve as a negative control.
  Interventions: Drug: Negative control

INTERVENTIONS:
Drug: GSK2894512 cream — GSK2894512 is a white to off-white cream that will be applied topically in 3 different concentrations (0.5% [5 milligram (mg)/gram (g)], 1% [10 mg/g], and 2% [20 mg/g]).
  Arms: GSK2894512 0.5%; GSK2894512 1%; GSK2894512 2%
Drug: Vehicle cream — Vehicle cream does not contain any active pharmaceutical ingredient.
  Arms: Vehicle
Drug: Positive control — Positive control contains sodium lauryl sulfate solution 0.1% (1 mg/g).
  Arms: Sodium lauryl sulfate 0.1%
Drug: Negative control — Negative control contains petrolatum.
  Arms: Petrolatum

SUMMARY:
This study is conducted to assess the potential of topically-applied GSK2894512 cream at 3 concentrations (0.5%, 1%, and 2%) to induce skin irritation at the site of application in healthy subjects. Results from this study will be considered when selecting the concentration(s) of GSK2894512 to evaluate in the Phase II and Phase III clinical safety and efficacy studies. Approximately 40 subjects will be enrolled in order to have at least 30 evaluable subjects complete the study. The total duration of subject participation may be up to 50 days.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years, inclusive, at time of consent.
* In generally good overall health with healthy skin in the potential test sites on the back.
* Skin tone in the potential test sites on the back such that erythema and other dermal reactions can be easily visualized, i.e., Fitzpatrick skin types I (always burns; never tans), II (usually burns; tans with difficulty), III (sometimes mild burn; gradually tans), or IV (rarely burns; tans with ease). Determination of skin types is based on sunburn and tanning history in response to the first 30 to 45 minutes of sun exposure.
* A woman is eligible to participate if she is of non-childbearing potential, defined as a woman with functioning ovaries who has a documented bilateral tubal ligation/sterilization or hysterectomy, bilateral oopherectomy, or postmenopausal with at least 12 months of spontaneous amenorrhea.

Exclusion Criteria:

* History of known or suspected intolerance to GSK2894512, any of the ingredients of the study products, adhesive tape/plaster, or the test chambers.
* Inability to evaluate the skin at and around the potential test sites on the back due to sunburns, unevenness in skin tone, tattoos, scars, excessive hair, freckles, birthmarks, moles, or other skin damage or abnormality.
* Clinically-relevant skin disease, including psoriasis, eczema, atopic dermatitis, acne, dysplastic nevi, or other skin pathologies, or a history of skin cancer, that may, in the opinion of the investigator, contraindicate participation or interfere with test site evaluations.
* Considered immunocompromised, or has a clinically-relevant history of or currently suffering from any disease or condition that, in the opinion of the investigator, might affect the evaluation of the study product or place the subject at undue risk.
* Used prohibited concomitant medications or products within the defined washout periods before the Day 1 visit. This includes investigational products, allergy injections, immunizations, corticosteroids, immunomodulators, anti-inflammatories, antihistamines, selective leukotriene receptor antagonists, mast cell stabilizers, and topical medications or products at and around the potential test sites.
* Participation in any interventional clinical study within 4 weeks of the Day 1 Visit.
* A clinically relevant history of or current evidence of abuse of alcohol or other drugs.
* Considered vulnerable (e.g., individuals in detention/institutionalized due to legal or regulatory order).
* Employee of the study center, bioskin GmbH, Parexel, GlaxoSmithKline (GSK), or Stiefel who is involved in the study, or an immediate family member (e.g., partner, offspring, parents, siblings, or sibling's offspring) of an employee who is involved in the study.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). Alanine aminotransferase (ALT), alkaline phosphatase, or bilirubin >1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%).
* QTc >=450 millisecond (msec) or QTc >=480 msec for subjects with bundle branch block. The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF), with machine overread. The QTc should be based on single or averaged QTc values of triplicate ECGs obtained over a brief recording period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2014-07-02 (Actual); Study Completion 2014-07-02 (Actual)

PRIMARY OUTCOMES:
Mean cumulative irritation score | 21 Days
  It is the sum of dermal response irritation scores from Day 2 through Day 22 divided by the number of non-missing observations
Total cumulative irritation score | 21 Days
  It is the sum of dermal response irritation scores from Day 2 through Day 22

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) and treatment-related AEs | Up to Day 22
  All AEs and serious adverse events will be collected from the time a subject consents to participate in the study through the final study visit
Change from baseline in vital signs | Screening, Day 1, Day 2, Day 4, Day 6, Day 8, Day 10, Day 12, Day 14, Day 16, Day 18, Day 20 and Day 22
  Vital signs include heart rate, blood pressure, and oral temperature
Change from baseline in clinical laboratory parameters | Screening, Day 11 (+/-2 days) and Day 22
  Laboratory parameters include haematology and, clinical chemistry tests
Change from baseline in electrocardiogram (ECG) findings | Screening, Day 11 (+/-2 days) and Day 22 (+/-2 days)
  Single 12-lead ECGs will be obtained using an ECG machine to monitor cardiac safety
Plasma trough concentrations of GSK2894512 | Day 11 (+/- 2 days) and Day 22
  Trough concentration is the minimum concentration of GSK2894512 observed after its administration and just prior to the administration of a subsequent dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Baltimore, Maryland, United States
- GSK Investigational Site, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 117191 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/117191?search=study&search_terms=117191#rs
- Available data/document: Study Protocol: 117191 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117191 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117191 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117191 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 117191 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117191 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register